CLINICAL TRIAL: NCT04097184
Title: Efficacy of Dorso-lateral Prefrontal Cortex Stimulation by tDCS in Patients With Motor Conversion Disorder - Multicentre Randomized Double Blind Assay
Brief Title: Efficacy of Dorso-lateral Prefrontal Cortex Stimulation by tDCS in Motor Conversion Disorder Patients
Acronym: CONVERSTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRC-N/2018/IC-01
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Conversion Disorder
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Intervention Model Description: Prospective multicentre controlled randomized, double-blind, two-arm study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will then be randomized and assigned to one of the 2 groups: the first group will receive a series of 10 effective stimulation sessions (experimental group "active tDCS") and the second group will receive a series of 10 placebo stimulation sessions (control group "sham tDCS").
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "active tDCS" group (Active Comparator): Patients will benefit from a series of 10 double-blind effective tDCS stimulation sessions over a period of 5 days (Monday to Friday): each stimulation series will include two daily stimulation sessions spaced 3 hours apart for 5 days.
  Interventions: Device: Neurostimulation with non-implanted electrodes
- "sham tDCS" group (Sham Comparator): Patients will benefit from a series of 10 double-blind placebo tDCS stimulation sessions over a period of 5 days (Monday to Friday): each stimulation series will include two daily stimulation sessions spaced 3 hours apart for 5 days.
  Interventions: Device: Neurostimulation with non-implanted electrodes

INTERVENTIONS:
Device: Neurostimulation with non-implanted electrodes — Neurostimulation with non-implanted electrodes

SUMMARY:
Conversion disorder refers to impaired voluntary motor or sensory functions that are not compatible with a well-known neurological condition. This disorder affects up to 30% of hospitalized patients in neurology departments and symptoms persist in 35% of patients after 12 years of evolution. Despite a poor prognosis, no treatments have been validated to date.

The development of non-invasive brain stimulation techniques has allowed the creation of treatments focused on dysfunctional brain regions associated with motor conversion disorder. Hypoactivation of prefrontal dorso-lateral cortex underlies the course of functional motor symptoms. Results of the HYCORE study conducted at Nîmes University Hospital (including 20 patients, clinicaltrial.gov NCT02329626) confirmed these results and related hypoactivation of PFDLC to persistent motor disability at 3 months and 6 months follow-up. Activation of the PFDLC could restore executive control and thus promote the recovery of motor symptoms.

However, in most repeated Transcranial Magnetic Stimulation (rTMS) the primary motor areas were targeted and the clinical improvement was related to self-suggestion induced by the motor response produced.

Among the different techniques, transcranial Direct Current Stimulation (tDCS) is a medical neuromodulation device that delivers a direct, low-intensity electric current to cortical areas, facilitating neuronal activity. Recently, PFDLC stimulation via tDCS has been used to treat several neuropsychiatric disorders and shown to be effective in depression. In addition, this technique has several advantages compared to rTMS: its use is simpler and costs 5 to 8 times less, the device is portable and there is no titration procedure. The tolerance of the tDCS is also better with no risk of epileptic seizure, neuronal depolarization being absent.

DETAILED DESCRIPTION:
Conversion disorder, also called "functional neurological disorder" (DSM-5), refers to impaired voluntary motor or sensory functions that are not compatible with a well-known neurological condition. This disorder affects up to 30% of hospitalized patients in neurology departments (Carson et al. 2000) and the symptoms persist in 35% of patients after 12 years of evolution (Stone et al. 2003). Despite a poor prognosis, no treatments have been validated to date.

The development of non-invasive brain stimulation techniques has allowed the creation of focused treatments on dysfunctional brain regions associated with motor conversion disorder. A hypoactivation of prefrontal dorso-lateral cortex (PFDLC) underlies the course of functional motor symptoms (Spence et al. 2000); (Voon et al.2011); (Conejero et al. 2017). Results of the HYCORE study that the investigators conducted at Nîmes University Hospital (including 20 patients, clinicaltrial.gov NCT02329626) confirmed these results and related hypoactivation of PFDLC to persistent motor disability at 3 months and 6 months follow-up. Activation of the PFDLC could restore executive control and thus promote the recovery of motor symptoms.

However, in the majority of repeated Transcranial Magnetic Stimulation (rTMS) the primary motor areas were targeted (Pollak et al. 2014) and the clinical improvement was related to self-suggestion induced by the motor response produced.

Among the different techniques, transcranial Direct Current Stimulation (tDCS) is a medical neuromodulation device that delivers a direct, low-intensity electric current to cortical areas, facilitating neuronal activity. Recently, PFDLC stimulation via tDCS has been used to treat several neuropsychiatric disorders and shown to be effective in depression. In addition, this technique has several advantages compared to rTMS: its use is simpler and costs 5 to 8 times less, the device is portable and there is no titration procedure. The tolerance of the tDCS is also better with no risk of epileptic seizure, neuronal depolarization being absent.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent.
* The patient is at least (≥) 18 years old and 65 years old at the most (≤). The risk of an increased frequency of somatic comorbidity, drug co-prescription, and cognitive impairment prompts us to limit recruitment to age 65 in this study.
* The patient is hospitalized or followed in consultation.
* Patient is available for a follow-up of 6 months.
* With current DSM-5 criteria for conversion disorder during more than 10 days, motor type (i.e. with paralysis or motor weakness) and initial EDSS score ≥ 3 or initial WHO Score is ≥ 2

Exclusion Criteria:

* The patient is participating in another interventional trial.
* The patient refuses to sign the consent.
* It is impossible to correctly inform the patient.
* The patient is pregnant or breastfeeding.
* Specialized neurological clinical examination and the performing of brain and medullary MRI reveal an organic neurological involvement.
* Current episode of mania, hypomania, diagnosis of substance abuse/dependence (excluding smoking), diagnosis of schizophrenia over lifetime, severe neurological pathology (epilepsy, stroke, brain tumor).
* Patient with a contraindication to MRI (for patients enrolled in Nîmes).
* Acute eczema at the electrodes loci.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of tDCS stimulation of the left PFDLC to treat motor disability in patients with conversion disorder 3 months after the intervention. | 3 months after the intervention
  Evaluation of the efficacy of tDCS stimulation of the left PFDLC to treat motor disability in patients with conversion disorder at 3 months after the stimulation procedure with the EDSS (Expanded Disability Status Scale). The Expanded Disability Status Scale is a rating scale of disability divided into eight systems or functional parameters, four major:
  pyramidal function, cerebellar function, sensory function and brainstem function; four minor: sphincters,vision, mind and others. An encrypted score of increasing severities (0 to 6 or 7) is given to each functional parameter. The overall score of the scale is measured on a scale of 20 levels (0 to 10 per half-point). Up to level 3.5, the score obtained in each functional parameter and the number of affected functional parameters automaticaly determines the EDSS score.
  From 4 to 7, the definition of each level is also given by the inability to walk (ability to walk without stopping - need for assistance).

SECONDARY OUTCOMES:
Evaluation of the efficacy on motor symptoms at D7 with NIHSS | 7 days after the intervention
  Evaluation of the efficacy on motor symptoms at Day 7 with the National Institute of Health Stroke Score (NIHSS). The National Institute of Health Stroke Score includes the following domains : level of consciousness, eye movements, integrity of visual fields, facial movements, arm and leg muscle strength, sensation, coordination, language, speech and neglect. Each impairment is scored on an ordinal scale ranging from 0 to 2, 0 to 3, or 0 to 4. Item scores are summed to a total score ranging from 0 to 42 (the higher the score, the more severe the stroke). Duration = 10 minutes
Evaluation of the persistence of efficacy on motor symptoms at 1 month | 1 month after the intervention
  Evaluation of the efficacy on motor symptoms at 1 month with National Institute of Health Stroke Score (NIHSS). The National Institute of Health Stroke Score includes the following domains : level of consciousness, eye movements, integrity of visual fields, facial movements, arm and leg muscle strength, sensation, coordination, language, speech and neglect. Each impairment is scored on an ordinal scale ranging from 0 to 2, 0 to 3, or 0 to 4. Item scores are summed to a total score ranging from 0 to 42 (the higher the score, the more severe the stroke). Duration = 10 minutes
Evaluation of the persistence of efficacy on motor symptoms at 3 months | 3 months after the intervention
  Evaluation of the efficacy on motor symptoms at 3 months with the National Institute of Health Stroke Score (NIHSS). The National Institute of Health Stroke Score includes the following domains : level of consciousness, eye movements, integrity of visual fields, facial movements, arm and leg muscle strength, sensation, coordination, language, speech and neglect. Each impairment is scored on an ordinal scale ranging from 0 to 2, 0 to 3, or 0 to 4. Item scores are summed to a total score ranging from 0 to 42 (the higher the score, the more severe the stroke). Duration = 10 minutes
Evaluation of the persistence of efficacy on motor symptoms at 6 months | 6 months after the intervention
  Evaluation of the efficacy on motor symptoms at 6 months with National Institute of Health Stroke Score (NIHSS). The National Institute of Health Stroke Score includes the following domains : level of consciousness, eye movements, integrity of visual fields, facial movements, arm and leg muscle strength, sensation, coordination, language, speech and neglect. Each impairment is scored on an ordinal scale ranging from 0 to 2, 0 to 3, or 0 to 4. Item scores are summed to a total score ranging from 0 to 42 (the higher the score, the more severe the stroke). Duration = 10 minutes
Evaluation of the efficacy on motor disability with EDSS score at D7. | 7 days after the intervention
  Evaluation of the efficacy of the intervention on motor symptoms at D7 using the Expanded Disability Status Scale (EDSS). The Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis. The scale was developed by John F. Kurtzke and an EDSS calculator is available on line. The EDSS is based on a neurological examination by a clinician, however a number of versions have been developed to enable patient self-administration.The EDSS quantifies disability in eight Functional Systems (FS) by assigning a Functional System Score (FSS) in each of these functional systems: pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral,other. The scale ranges from 0.0 (normal neurological examination) to 10.0 (death due to multiple sclerosis).
Evaluation of the persistence of efficacy on motor disability with EDSS at 1 month | 1 month after the intervention
  Evaluation of the persistence of efficacy of the intervention using the Expanded Disability Status Scale (EDSS) at 1 month. The Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis. The scale was developed by John F. Kurtzke and an EDSS calculator is available on line. The EDSS is based on a neurological examination by a clinician, however a number of versions have been developed to enable patient self-administration.The EDSS quantifies disability in eight Functional Systems (FS) by assigning a Functional System Score (FSS) in each of these functional systems: pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral,other. The scale ranges from 0.0 (normal neurological examination) to 10.0 (death due to multiple sclerosis).
Evaluation of the persistence of efficacy on motor disability with EDSS at 6 months. | 6 month after the intervention
  Evaluation of the persistence of efficacy of the intervention on motor disability using the Expanded Disability Status Scale (EDSS) at 6 months.The Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis. The scale was developed by John F. Kurtzke and an EDSS calculator is available on line. The EDSS is based on a neurological examination by a clinician, however a number of versions have been developed to enable patient self-administration.The EDSS quantifies disability in eight Functional Systems (FS) by assigning a Functional System Score (FSS) in each of these functional systems: pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral,other. The scale ranges from 0.0 (normal neurological examination) to 10.0 (death due to multiple sclerosis).
WHO score at D7 | 7 days after the intervention
  Evaluation of the efficacy of the intervention on motor disability with WHO Performance Status at Day 7. The WHO (World Health Organization) Performance Status is a 5-point scale and is the simplest and fastest indicator to judge the state of autonomy of a person:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
WHO score at 1 month | 1 month after the intervention
  Evaluation of the persistence of efficacy of the intervention on motor disability with WHO score at 1 month.The WHO (World Health Organization) Performance Status is a 5-point scale and is the simplest and fastest indicator to judge the state of autonomy of a person:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
WHO score at 3 months | 3 months after the intervention
  Evaluation of the persistence of efficacy of the intervention on motor disability with WHO at 3 months.The WHO (World Health Organization) Performance Status is a 5-point scale and is the simplest and fastest indicator to judge the state of autonomy of a person:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
WHO score at 6 months | 3 months after the intervention
  Evaluation of the persistence of efficacy of the intervention on motor disability with WHO at 3 months. The WHO (World Health Organization) Performance Status is a 5-point scale and is the simplest and fastest indicator to judge the state of autonomy of a person:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair
  5. Dead
CGI (Clinical Global Impression) scores at Day 7 | 7 days after the intervention
  Evaluation of the efficacy on motor disability with Clinical Global Impression score at Day 7. The CGI is a set of two scales with points ranging from 1 -7.
  The first set describes the Severity of Illness ( 1 = no illness or symptoms of disorder for the past 7 days and 7 = among the most drastically ill patients) The second set describes the Global Improvement (1 = very much improved, 7 = very much worse)
CGI (Clinical Global Impression) score at 3 months | 3 months after the intervention
  Evaluation of the persistence of efficacy of the intervention on motor disability with Clinical Global Impression scores at 3 months. The CGI is a set of two scales with points ranging from 1 -7.
  The first set describes the Severity of Illness ( 1 = no illness or symptoms of disorder for the past 7 days and 7 = among the most drastically ill patients) The second set describes the Global Improvement (1 = very much improved, 7 = very much worse)
CGI (Clinical Global Impression) score at 6 months | 6 months after the intervention
  Evaluation of the persistence of efficacy of the intervention on motor disability with Clinical Global Impression scores at 6 months. The CGI is a set of two scales with points ranging from 1 -7.
  The first set describes the Severity of Illness ( 1 = no illness or symptoms of disorder for the past 7 days and 7 = among the most drastically ill patients) The second set describes the Global Improvement (1 = very much improved, 7 = very much worse)
Modified Rankin (mRS) score at D7 | 7 days after the intervention
  Evaluation of the efficacy on motor disability with modified Rankin (mRS) scores at D7 months. The Modified Rankin (mRS) score is a scale ranging from 0 - 6 with 0 being no symptoms at all. 3 = moderate disability despite symptoms but able to walk without asistance and 6 = dead.
Modified Rankin (mRS) score at 1 month | 1 month after the intervention
  Evaluation of the efficacy on motor disability with modified Rankin (mRS) scores at 1 month. The Modified Rankin (mRS) score is a scale ranging from 0 - 6 with 0 being no symptoms at all. 3 = moderate disability despite symptoms but able to walk without asistance and 6 = dead.
Modified Rankin (mRS) score at 3 months | 3 months after the intervention
  Evaluation of the efficacy on motor disability with modified Rankin (mRS) scores at 1 month.The Modified Rankin (mRS) score is a scale ranging from 0 - 6 with 0 being no symptoms at all. 3 = moderate disability despite symptoms but able to walk without asistance and 6 = dead.
Modified Rankin (mRS) score at 6 months | 6 months after the intervention
  Evaluation of the efficacy on motor disability with modified Rankin (mRS) score at 6 months. The Modified Rankin (mRS) score is a scale ranging from 0 - 6 with 0 being no symptoms at all. 3 = moderate disability despite symptoms but able to walk without asistance and 6 = dead.
Evaluation of disability related to abnormal movements - CGI at D7. | 7 days after the intervention
  Evaluate the efficacy on disability related to abnormal movements with Clinical Global Impression scores at Day 7.The CGI is a set of two scales with points ranging from 1 -7.
  The first set describes the Severity of Illness ( 1 = no illness or symptoms of disorder for the past 7 days and 7 = among the most drastically ill patients) The second set describes the Global Improvement (1 = very much improved, 7 = very much worse)
Evaluation of disability related to abnormal movements - CGI at 1 month. | 1 month after the intervention
  Evaluate the persistence of efficacy on disability related to abnormal movements with Clinical Global Impression scores at 1 month.The CGI is a set of two scales with points ranging from 1 -7.
  The first set describes the Severity of Illness ( 1 = no illness or symptoms of disorder for the past 7 days and 7 = among the most drastically ill patients) The second set describes the Global Improvement (1 = very much improved, 7 = very much worse)
Evaluation of disability related to abnormal movements - CGI at 3 months. | 3 months after the intervention
  Evaluate the persistence of efficacy on disability related to abnormal movements with Clinical Global Impression scores at 3 months. The CGI is a set of two scales with points ranging from 1 -7.
  The first set describes the Severity of Illness ( 1 = no illness or symptoms of disorder for the past 7 days and 7 = among the most drastically ill patients) The second set describes the Global Improvement (1 = very much improved, 7 = very much worse)
Evaluation of disability related to abnormal movements - CGI at 6 months. | 6 months after the intervention
  Evaluation of the persistence of efficacy on disability related to abnormal movements with Clinical Global Impression scores at 6 months. The CGI is a set of two scales with points ranging from 1 -7.
  The first set describes the Severity of Illness ( 1 = no illness or symptoms of disorder for the past 7 days and 7 = among the most drastically ill patients) The second set describes the Global Improvement (1 = very much improved, 7 = very much worse)
Efficacy on depression and anxiety level assessed with the HAD score (HADS) at D7 | 7 days after the intervention
  Evaluation of the efficacy of the intervention on depression and anxiety level with the Hospital Anxiety and Depression Scale (HADS) at D7. The Hospital Anxiety and Depression Scale (HADS) questionnaire (Zigmond and Snaith 1983) validated in French (Lépine et al., 1985) is commonly used in screening for anxio-depressive disorders in studies; it is The HADS questionnaire consists of 14 questions (7 questions about anxiety and 7 questions about depression). Each question is an MCQ with four possible answers. The final score gives a ranking of anxiety and depressive symptoms as follows:
  * 0-7: normal
  * 8-10: average
  * 11-14: moderate
  * 15 to 21: severe This scale is used in this study to characterize the state of anxiety of the population and therefore for descriptive purposes.
Efficacy on depression and anxiety level assessed with the HAD score (HADS) at 1 month | 1 month after the intervention
  Evaluation of the persistence of efficacy on depression and anxiety level with the Hospital Anxiety and Depression Scale (HADS) at 1 month. The Hospital Anxiety and Depression Scale (HADS) questionnaire (Zigmond and Snaith 1983) validated in French (Lépine et al., 1985) is commonly used in screening for anxio-depressive disorders in studies; it is The HADS questionnaire consists of 14 questions (7 questions about anxiety and 7 questions about depression). Each question is an MCQ with four possible answers. The final score gives a ranking of anxiety and depressive symptoms as follows:
  * 0-7: normal
  * 8-10: average
  * 11-14: moderate
  * 15 to 21: severe This scale is used in this study to characterize the state of anxiety of the population and therefore for descriptive purposes.
Efficacy on depression and anxiety level assessed with the HAD score (HADS) at 3 months . | 3 months after the intervention
  Evaluation of the persistence of efficacy on depression and anxiety level assessed with the Hospital Anxiety and Depression Scale (HADS) at D7 and persistence at 3 months.The Hospital Anxiety and Depression Scale (HADS) questionnaire (Zigmond and Snaith 1983) validated in French (Lépine et al., 1985) is commonly used in screening for anxio-depressive disorders in studies; it is The HADS questionnaire consists of 14 questions (7 questions about anxiety and 7 questions about depression). Each question is an MCQ with four possible answers. The final score gives a ranking of anxiety and depressive symptoms as follows:
  * 0-7: normal
  * 8-10: average
  * 11-14: moderate
  * 15 to 21: severe This scale is used in this study to characterize the state of anxiety of the population and therefore for descriptive purposes.
Efficacy on depression and anxiety level assessed with the HAD score (HADS) at 6 months. | 6 months after the intervention
  Evaluation of the persistence of efficacy on depression and anxiety level assessed with the HAD score (HADS) at 6 months.The Hospital Anxiety and Depression Scale (HADS) questionnaire (Zigmond and Snaith 1983) validated in French (Lépine et al., 1985) is commonly used in screening for anxio-depressive disorders in studies; it is The HADS questionnaire consists of 14 questions (7 questions about anxiety and 7 questions about depression). Each question is an MCQ with four possible answers. The final score gives a ranking of anxiety and depressive symptoms as follows:
  * 0-7: normal
  * 8-10: average
  * 11-14: moderate
  * 15 to 21: severe This scale is used in this study to characterize the state of anxiety of the population and therefore for descriptive purposes.
Interaction between time from symptom onset to inclusion in the study, initial severity of abnormal movements and efficacy of motor symptom treatment measured with EDSS at D7 | 7 days after the intervention
  Evaluation of the interaction between time from symptom onset to inclusion in the study, the initial severity of abnormal movements and the efficacy of motor symptom treatment measured with EDSS at D7.
Interaction between time from symptom onset to inclusion in the study, initial severity of abnormal movements and efficacy of motor symptom treatment measured with EDSS at 1 month | 1 month after the intervention
  Evaluation of the interaction between time from symptom onset to inclusion in the study, the initial severity of abnormal movements and the efficacy of motor symptom treatment measured with EDSS at 1 month.
Interaction between time from symptom onset to inclusion in the study, initial severity of abnormal movements and efficacy of motor symptom treatment measured with EDSS at 3 months | 3 months after the intervention
  Evaluation of the interaction between time from symptom onset to inclusion in the study, the initial severity of abnormal movements and the efficacy of motor symptom treatment measured with EDSS at 3 months.
Interaction between time from symptom onset to inclusion in the study, initial severity of abnormal movements and efficacy of motor symptom treatment measured with EDSS at 6 months | 6 months after the intervention
  Evaluation of the interaction between time from symptom onset to inclusion in the study, the initial severity of abnormal movements and the efficacy of motor symptom treatment measured with EDSS at 6 months.
Tolerance to tDCS stimulation D2 - D6 Brunoni | From 2 days to 6 days after the intervention
  Evaluate the tolerance to tDCS stimulation sessions from D2 to D6 with Brunoni's questionnaire.To monitor and evaluate the potential adverse effects of tDCS in patients receiving this treatment, Brunoni et al. (2011) proposed a structured questionnaire. The patient answers questions regarding symptoms or side-effects on different parts of the body and their severity ranges from 1 - 4 (1 = absent, 2 = mild, 3 = moderate, 4 = severe). The probability of these symptoms or side-effects being related to the tDCS stimulation treatment is also noted from 1 - 5 ( 1 = none, 2 = remote, 3 = possible, 4 = probable, 5 = definite).
Correlation between putative modification of motor symptoms and changes in activity (rest / motor imagery task) of the PFDLC monitored by brain fMRI at Day 0 and Day 7. | Day 0 and Day 7
  Evaluation of the correlation between putative modification of motor symptoms and changes in activity (at rest or during a motor imagery task) of the PFDLC monitored by functional brain MRI at day 0 and day 7, i.e. search for early response markers to the treatment.
Evaluation of Dissociative Experiences Scale | 7 days after the intervention
  Evaluate the influence of the initial level of psychic dissociation assessed with the DES scale at D0 on the efficacy of tDCS treatment on the motor's symptoms of CD at day 7
Evaluation of Dissociative Experiences Scale | 1 month after the intervention
  Evaluate the influence of the initial level of psychic dissociation assessed with the DES scale at D0 on the efficacy of tDCS treatment on the motor's symptoms of CD
Evaluation of Dissociative Experiences Scale | 3 month after the intervention
  Evaluate the influence of the initial level of psychic dissociation assessed with the DES scale at D0 on the efficacy of tDCS treatment on the motor's symptoms of CD
Evaluation of Dissociative Experiences Scale | 6 month after the intervention
  Evaluate the influence of the initial level of psychic dissociation assessed with the DES scale at D0 on the efficacy of tDCS treatment on the motor's symptoms of CD
Evaluate the evolution of dissociation Experiences Scale | 7 days after the intervention
  Evaluate the influence of the initial level of psychic dissociation assessed with the DES scale at D0 on the efficacy of tDCS treatment on the motor's symptoms of CD
Evaluate the evolution of dissociation Experiences Scale | 1 month after the intervention
  Evaluate the influence of the initial level of psychic dissociation assessed with the DES scale at D0 on the efficacy of tDCS treatment on the motor's symptoms of CD
Evaluate the evolution of dissociation Experiences Scale | 3 month after the intervention
  Evaluate the influence of the initial level of psychic dissociation assessed with the DES scale at D0 on the efficacy of tDCS treatment on the motor's symptoms of CD
Evaluate the evolution of dissociation Experiences Scale | 6 month after the intervention
  Evaluate the influence of the initial level of psychic dissociation assessed with the DES scale at D0 on the efficacy of tDCS treatment on the motor's symptoms of CD
Evaluate the concordance of the CGI scale between the neurologist's assessment and the psychiatrist's assessment. | 7 days after the intervention
  Score at the CGI questionnaire
Evaluate the concordance of the CGI scale between the neurologist's assessment and the psychiatrist's assessment. | 1 month after the intervention
  Score at the CGI questionnaire
Evaluate the concordance of the CGI scale between the neurologist's assessment and the psychiatrist's assessment. | 3 month after the intervention
  Score at the CGI questionnaire
Evaluate the concordance of the CGI scale between the neurologist's assessment and the psychiatrist's assessment. | 6 month after the intervention
  Score at the CGI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ismael CONEJERO, Dr., Principal Investigator — CHU de Nîmes (Nîmes University Hospital)
Locations (8):
- France (8):
  - Centre Hospitalier Universitaire, Nîmes, Gard
  - Hôpital La Colombière Service de Psychiatrie, Montpellier, Hérault
  - CHU de Montpellier Hôpital Gui De Chauliac Service de Neurologie, Montpellier, Hérault
  - Hôpital Lapeyronie, Montpellier, Hérault
  - Hospices Civils de Lyon Hôpital Edouard Herriot, Lyon
  - CHU de Nantes, Nantes
  - Clinique St Exupery, Toulouse
  - Hôpital Saint-Antoine Service de Psychiatrie APHP, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No